CLINICAL TRIAL: NCT03587584
Title: Comparing Liposomal Bupivacaine to Bupivacaine Interscalene Blocks for Arthroscopic Rotator Cuff Repair Surgery: A Randomized Controlled Trial
Brief Title: Liposomal Bupivacaine Interscalene Blocks for Rotator Cuff Repair
Acronym: RCR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANES-2018-26660
Record Dates: First submitted 2018-06-20; First posted 2018-07-16 (Actual); Results first posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- liposomal bupivacaine (Experimental): These patients receive an interscalene block with liposomal bupivacaine.
  Interventions: Drug: liposomal bupivacaine
- bupivacaine (Active Comparator): These patients receive an interscalene block with bupivacaine.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: liposomal bupivacaine — Experimental
  Arms: liposomal bupivacaine
Drug: Bupivacaine — Active Comparator
  Arms: bupivacaine

SUMMARY:
The purpose of this study is to compare pain control after arthroscopic rotator cuff repair surgery using either liposomal bupivacaine or bupivacaine when injected in an interscalene block. Both medications, liposomal bupivacaine and bupivacaine, are standard of care in these types of surgeries.

DETAILED DESCRIPTION:
All patients will receive preoperative oral multimodal medications consisting of acetaminophen 975 mg, gabapentin 300 mg, and Celebrex 400 mg.

After completion of the preoperative process the patient will be placed in the supine position with the head of the bed elevated 30 degrees with standard ASA monitors applied. Sedation will be provided with midazolam 0-2 mg and propofol 50 mg. The interscalene groove will be identified with the ultrasound. Using sterile technique, a 21g Nerve block needle will then be inserted and advanced under ultrasound guidance until it is in the interscalene groove. Once in the interscalene, 20 mL of local anesthetic will be injected, with 10 mL deposited at the top of the brachial plexus and 10 mL at the bottom. In the study group, 5 mL of each 0.5% bupivacaine and LB will be injected at each location. The control group with have 20 mL of 0.5% bupivacaine divided between the injection sites. The patient will be monitored in the preoperative area until he/she is brought into the operating room for their procedure. A working block prior to surgery will be confirmed via sensory testing of the shoulder.

All patients will undergo a standard induction with propofol 1.5-3.0 mg/kg, ondansetron 4 mg, dexamethasone 10 mg and ketamine 0.25 mg/kg. A MAC or general with LMA or ETT will be placed and an opioid sparing technique will occur. Standardized maintenance will be a propofol infusion without neuromuscular blockers. 25-50 mcg of IV Fentanyl will be utilized for increases in heart rate greater than 20% or increases in systolic blood pressure above baseline.

Once in the operating room the surgeon will use 10 mL of 0.25% bupivacaine for skin, subcutaneous, and intraarticular injection.

When the operation is complete, the patient will be woken up and brought to the PACU. There the patient will receive IV fentanyl for a pain score of greater than 7. If more than 100 mcg of fentanyl is given and pain still remains above a 7 then IV hydromorphone will be used. A dose of 5-10 mg of oral oxycodone (or 2-4 mg of oral hydromorphone) will be given as soon as the patient is able to tolerate oral medication per standard protocol: If their pain score is 4-6 (on the Visual Analog Scale) then 5mg oral oxycodone (2 mg hydromorphone) can be administered, if their pain is between 7 to 10 then 10 mg of oxycodone (or 4 mg of hydromorphone) can be administered. Once the patient meets discharge criteria, they will be discharged home where each day they will fill out a pain diary. Additionally, a member of the research team will call the patient for signs of complications and ask the patient their current pain score, total opioid pills taken and non-opioid pain medication taken at 24, 48, and 72 hours postoperatively. Additionally, they will perform a Quality of Recovery Score survey at 72 hours, and 14 days postoperatively. An Ultrasound of the diaphragm will be completed by a blinded anesthesiologist in the PACU to assess diaphragm function.

All patients will be discharged with acetaminophen 975 mg q6 hours & ibuprofen 600 mg q6 hours, taken in intervals such that the patient is taking one of these medications every 3 hours. And then hydromorphone 2mg pills #60 dosing 1-2 pills q4 hours prn severe pain or oxycodone 5 mg pills #60 dosing 1-2 pills q 4 hours prn severe pain.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged greater than 18 years of age that are undergoing arthroscopic rotator cuff surgery

Exclusion Criteria:

* Patients with allergy to local anesthetics
* Patients with daily use of opioids for more than 3 weeks prior to surgery
* Patients who refuse
* Patients with coagulopathy
* Patients who are non-english speaking
* Patients who do not have access to a telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tenzin Desa, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Flaherty JM, Berg AA, Harrison A, Braman J, Pearson JM, Matelich B, Kaizer AM, Hutchins JL. Comparing liposomal bupivacaine plus bupivacaine to bupivacaine alone in interscalene blocks for rotator cuff repair surgery: a randomized clinical trial. Reg Anesth Pain Med. 2022 May;47(5):309-312. doi: 10.1136/rapm-2021-103349. Epub 2022 Feb 21. PMID 35190468

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liposomal Bupivacaine | Bupivacaine
Started | 37 | 42
Completed | 33 | 33
Not Completed | 4 | 9
Not completed — SOC deviations | 4 | 6
Not completed — Incomplete data | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine | Bupivacaine | Total
Number analyzed (Participants) | 37 | 42 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 36 | 66
  >=65 years | 7 | 6 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 26 | 48
  Male | 15 | 16 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Total Intraoperative Opioids Used
Description: Total amount of opioid medications used during surgery. Opioids normalized to total morphine equivalents.
Time Frame: through end of surgery
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Liposomal Bupivacaine | Bupivacaine
Number analyzed (Participants) | 33 | 33
mg
  Intraoperative Fentanyl (mg) | .1 [.1 to .1] | .1 [.05 to .1]
  Intraoperative MME (mg) | 30 [30 to 30] | 30 [15 to 30]
  Intraoperative hydromorphone (mg) | 0 [0 to 0] | 0 [0 to 0]
  Intraoperative ketamine | 0 [0 to 0] | 0 [0 to 0]
  Intraoperative ketorolac (mg) | 0 [0 to 30] | 0 [0 to 30]

ADVERSE EVENTS:
Time Frame: 72 hours
Arm/Group | Liposomal Bupivacaine | Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 6/33 | 6/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liposomal Bupivacaine (N=33) | Bupivacaine (N=33)
Nausea (Gastrointestinal disorders) | 5 (5) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT03587584/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT03587584/ICF_001.pdf